CLINICAL TRIAL: NCT01077271
Title: PMOS to Evaluate the Compliance to Synagis (Palivizumab) Under Daily Pediatrician´s Conditions in Premature Infants 33 - 35 wGA Over 3 Consecutive Respiratory Syncytial Virus (RSV) Seasons in Austria
Brief Title: Compliance to Synagis (Palivizumab) Under Daily Pediatrician´s Conditions in Premature Infants 33 - 35 wGA
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Collaborators: Assign Data Management and Biostatistics GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: P11-040
Record Dates: First submitted 2010-02-25; First posted 2010-03-01 (Estimated); Results first posted 2012-08-21 (Estimated); Last update posted 2012-08-21 (Estimated); Status verified 2012-08

CONDITIONS: Premature Infants
Keywords: Premature infants; Respiratory Syncytial Virus (RSV); Compliance; Palivizumab
MeSH Terms: conditions — Premature Birth; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Premature infants 33 - 35 wGA prophylaxed with palivizumab: Premature infants 33 - 35 weeks gestational age (wGA) prophylaxed with Synagis (palivizumab)

SUMMARY:
Compliance to Synagis (palivizumab) is a key factor to obtain maximal protection against respiratory syncytial virus (RSV) infection as shown in the IMpact study. Many factors such as parents' knowledge of burden of respiratory syncytial virus disease or physicians' satisfaction with Synagis as well as the appropriate use of the product might influence compliance. The primary objective of this observational study is to evaluate the compliance to Synagis under daily pediatricians practice conditions in premature infants 33 to 35 weeks gestational age (wGA). Palivizumab, monoclonal antibody for passive immunoprophylaxis against severe respiratory syncytial virus disease, was administered according to usual clinical practice. Compliance was assessed using four criteria: The number of injections per participant per respiratory syncytial virus season, the body site where injections were administered, the interval in days between injections, and the dosage per administration. Originally the study was to include two respiratory syncytial virus seasons but was extended to a third season.

ELIGIBILITY:
Inclusion Criteria:

* Premature infant 33 to 35 weeks gestational age
* Younger than 3 months at respiratory syncytial virus season start
* At least 4 points according to the Austrian risk score according to Austrian guidelines: 1 point younger than 3 months (at start of respiratory syncytial virus season), 1 point neurologic disease, 1 point weight less than 10th percentile, 1 point discharge from hospital during respiratory syncytial virus season (1 Oct - 30 March), 1 point older siblings, 0.5 points multiple births, 0.5 points day care attendance, 0.5 points passive tobacco smoke exposure, 0.5 points socio-economic status (overcrowding)
* Synagis application (prescription)
* Signed authorization form for data use (parental authorization)

Exclusion Criteria:

* Patients without Synagis prescription
* Patients who meet contraindications as outlined in the latest version of Synagis summary of product characteristics (SmPC):

  * Patients with known hypersensitivity to palivizumab or any component of the formulation or other humanized monoclonal antibodies
* Patients with chronic lung disease
* Patients with congenital heart disease
* Greater than 36 weeks gestational age

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Medical practices specialized in pediatrics.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2008-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Astrid Dworan-Timler, MD, Study Director — Abbott Austria
Locations (45):
- Austria (45):
  - Site Reference ID/Investigator# 27772, Amstetten
  - Site Reference ID/Investigator# 52871, Amstetten
  - Site Reference ID/Investigator# 52873, Feldkirch
  - Site Reference ID/Investigator# 40437, Gänserndorf
  - Site Reference ID/Investigator# 30843, Hollabrunn
  - Site Reference ID/Investigator# 27767, Judenburg
  - Site Reference ID/Investigator# 27770, Klagenfurt
  - Site Reference ID/Investigator# 27777, Klosterneuburg
  - Site Reference ID/Investigator# 30842, Krems
  - Site Reference ID/Investigator# 27771, Leonding
  - Site Reference ID/Investigator# 52867, Linz
  - Site Reference ID/Investigator# 58943, Linz
  - Site Reference ID/Investigator# 18603, Linz
  - Site Reference ID/Investigator# 40445, Linz
  - Site Reference ID/Investigator# 52874, Linz
  - Site Reference ID/Investigator# 52870, Mattersburg
  - Site Reference ID/Investigator# 48262, Neufeld
  - Site Reference ID/Investigator# 27775, Purkersdorf
  - Site Reference ID/Investigator# 30850, Sankt Pölten
  - Site Reference ID/Investigator# 27765, Scheibbs
  - Site Reference ID/Investigator# 40440, Schörfling
  - Site Reference ID/Investigator# 27764, Telfs
  - Site Reference ID/Investigator# 40439, Traisen
  - Site Reference ID/Investigator# 30848, Tulln
  - Site Reference ID/Investigator# 27776, Tulln
  - Site Reference ID/Investigator# 30845, Vienna
  - Site Reference ID/Investigator# 30849, Vienna
  - Site Reference ID/Investigator# 40432, Vienna
  - Site Reference ID/Investigator# 40447, Vienna
  - Site Reference ID/Investigator# 27773, Vienna
  - Site Reference ID/Investigator# 52879, Vienna
  - Site Reference ID/Investigator# 27769, Vienna
  - Site Reference ID/Investigator# 40446, Vienna
  - Site Reference ID/Investigator# 52878, Vienna
  - Site Reference ID/Investigator# 27774, Vienna
  - Site Reference ID/Investigator# 27762, Vienna
  - Site Reference ID/Investigator# 27763, Vienna
  - Site Reference ID/Investigator# 40442, Vienna
  - Site Reference ID/Investigator# 30851, Vienna
  - Site Reference ID/Investigator# 58942, Vienna
  - Site Reference ID/Investigator# 30846, Vienna
  - Site Reference ID/Investigator# 30847, Vienna
  - Site Reference ID/Investigator# 57793, Vienna
  - Site Reference ID/Investigator# 30852, Vienna
  - Site Reference ID/Investigator# 40425, Vienna

REFERENCES:
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Premature Infants 33 - 35 wGA Prophylaxed With Palivizumab: Premature infants 33 - 35 weeks gestational age (wGA) prophylaxed with palivizumab
Period: Overall Study
Arm/Group | Premature Infants 33 - 35 wGA Prophylaxed With Palivizumab
Started | 124
Participants Treated With Palivizumab | 120
Number of Participants Analyzed | 120
Completed | 102
Not Completed | 22
Not completed — Parental desire | 8
Not completed — Screen failure, did not take palivizumab | 4
Not completed — Noncompliance | 2
Not completed — Quota used up (insurance reimb issue) | 2
Not completed — Changed doctors | 2
Not completed — Parents thought too many injections | 2
Not completed — End of RSV season nearly reached | 1
Not completed — Mother unconvinced of the necessity | 1

BASELINE CHARACTERISTICS:
Groups:
- RSV Season 1: Premature infants 33 - 35 weeks gestational age prophylaxed with palivizumab who were enrolled during the first respiratory syncytial virus season (01 Nov 2008 through 31 March 2009)
- RSV Season 2: Premature infants 33 - 35 weeks gestational age prophylaxed with palivizumab who were enrolled during the second respiratory syncytial virus season (01 Nov 2009 through 31 March 2010)
- RSV Season 3: Premature infants 33 - 35 weeks gestational age prophylaxed with palivizumab who were enrolled during the third respiratory syncytial virus season (01 Nov 2010 through 31 March 2011)
- No Matching RSV Season: Premature infants 33 - 35 weeks gestational age whose palivizumab administration did not occur within Season 1, 2 or 3
- Total: Total of all reporting groups
Arm/Group | RSV Season 1 | RSV Season 2 | RSV Season 3 | No Matching RSV Season | Total
Number analyzed (Participants) | 39 | 45 | 32 | 4 | 120
Age, Customized [Number; unit: Participants] — The chronological age of participants at study entry.
  Participants
    Less than 1 month | 1 | 1 | 2 | 1 | 5
    1 month | 10 | 15 | 7 | 0 | 32
    Greater than 1 and less than or equal to 2 months | 19 | 12 | 14 | 3 | 48
    3 months | 4 | 6 | 4 | 0 | 14
    4 to 4.5 months | 1 | 1 | 2 | 0 | 4
    5 months | 0 | 4 | 1 | 0 | 5
    6 months | 1 | 4 | 0 | 0 | 5
    7 months | 0 | 0 | 1 | 0 | 1
    8 months | 0 | 2 | 0 | 0 | 2
    9 months | 0 | 0 | 1 | 0 | 1
    10 months | 2 | 0 | 0 | 0 | 2
    Age not reported | 1 | 0 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 21 | 13 | 3 | 50
  Male | 26 | 24 | 19 | 1 | 70
Gestational age [Number; unit: Participants] — The gestational age of participants at birth in week of gestation.
  Participants
    23 weeks | 0 | 1 | 0 | 0 | 1
    28 weeks | 0 | 0 | 1 | 0 | 1
    31 weeks | 0 | 0 | 1 | 0 | 1
    33 weeks | 24 | 18 | 14 | 1 | 57
    34 weeks | 9 | 18 | 12 | 3 | 42
    35 weeks | 6 | 8 | 4 | 0 | 18
Body weight [Mean (Standard Deviation); unit: kilograms] — The body weight of participants at the first study visit.
  kilograms | 3.9 (1.4) | 3.8 (1.5) | 4.1 (1.6) | 3.5 (1.1) | 3.9 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Number of Injections Per Patient Per Season
Description: The average number of injections administered per participant within a respiratory syncytial virus season.
Time Frame: One RSV season (5 months)
Population: Participants who were administered palivizumab were included in the analysis.
Measure: Mean (Standard Deviation); unit: Injections administered
Groups:
- Total: Premature infants 33 - 35 weeks gestational age prophylaxed with palivizumab
Arm/Group | RSV Season 1 | RSV Season 2 | RSV Season 3 | No Matching RSV Season | Total
Number analyzed (Participants) | 39 | 45 | 32 | 4 | 120
Injections administered | 3.8 (1.3) | 3.9 (1.1) | 4.0 (1.4) | 1.0 (0.0) | 3.8 (1.3)

2. Primary Outcome: Body Site of Injections Per Administration
Description: The body site of injection administration for participants at each study visit.
Time Frame: One RSV season (5 months)
Population: The analysis population includes participants who were administered palivizumab and had data available for the study visits listed.
Measure: Number; unit: participants
Arm/Group | RSV Season 1 | RSV Season 2 | RSV Season 3 | No Matching RSV Season | Total
Number analyzed (Participants) | 39 | 45 | 32 | 4 | 120
participants
  Visit 1: Thigh | 38 | 44 | 29 | 4 | 115
  Visit 2: Thigh | 34 | 43 | 32 | 0 | 109
  Visit 3: Thigh | 31 | 42 | 23 | 0 | 96
  Visit 3: Other location | 0 | 0 | 1 | 0 | 1
  Visit 4: Thigh | 20 | 28 | 22 | 0 | 70
  Visit 4: Other location | 0 | 0 | 1 | 0 | 1
  Visit 5: Thigh | 15 | 13 | 15 | 0 | 43
  Visit 5: Other location | 0 | 0 | 1 | 0 | 1
  Visit 6: Thigh | 5 | 3 | 3 | 0 | 11
  Visit 6: Other location | 0 | 0 | 1 | 0 | 1
  Visit 7: Thigh | 2 | 3 | 0 | 0 | 5

3. Primary Outcome: Interval Between Administrations
Description: The average number of days that elapsed between palivizumab injections administered at the previous study visit.
Time Frame: One RSV season (5 months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Days
Groups:
- RSV Season 1 (S1): Premature infants 33 - 35 weeks gestational age prophylaxed with palivizumab who were enrolled during the first respiratory syncytial virus season (01 Nov 2008 through 31 March 2009)
- RSV Season 2 (S2): Premature infants 33 - 35 weeks gestational age prophylaxed with palivizumab who were enrolled during the second respiratory syncytial virus season (01 Nov 2009 through 31 March 2010)
- RSV Season 3 (S3): Premature infants 33 - 35 weeks gestational age prophylaxed with palivizumab who were enrolled during the third respiratory syncytial virus season (01 Nov 2010 through 31 March 2011)
- No Matching RSV Season (NS): Premature infants 33 - 35 weeks gestational age whose palivizumab administration did not occur within Season 1, 2 or 3
Arm/Group | RSV Season 1 (S1) | RSV Season 2 (S2) | RSV Season 3 (S3) | No Matching RSV Season (NS) | Total
Number analyzed (Participants) | 39 | 45 | 32 | 4 | 120
Days
  V2 (S1 n=33; S2 n=42; S3 n=29; NS n=0) | 28.5 (9.1) | 30.6 (9.2) | 28.6 (9.2) | NA (NA) — No data reported for this subgroup at this time point. | 29.4 (9.1)
  V3 (S1 n=32; S2 n=42; S3 n=24; NS n=0) | 33.2 (12.4) | 34.7 (12.1) | 30.3 (4.8) | NA (NA) — No data reported for this subgroup at this time point. | 33.1 (10.9)
  V4 (S1 n=20; S2 n=28; S3 n=23; NS n=0) | 34.5 (9.4) | 41.8 (48.2) | 32.0 (5.5) | NA (NA) — No data reported for this subgroup at this time point. | 36.6 (30.8)
  V5 (S1 n=15; S2 n=13; S3 n=16; NS n=0) | 33.4 (13.9) | 32.5 (12.9) | 28.4 (5.5) | NA (NA) — No data reported for this subgroup at this time point. | 31.3 (11.2)
  V6 (S1 n=6; S2 n=3; S3 n=4; NS n=0) | 24.8 (10.3) | 30.0 (1.7) | 29.5 (1.7) | NA (NA) — No data reported for this subgroup at this time point. | 27.5 (7.2)
  V7 (S1 n=2; S2 n=3; S3 n=0; NS n=0) | 34.0 (0.0) | 30.0 (1.7) | NA (NA) — No data reported for this subgroup at this time point. | NA (NA) — No data reported for this subgroup at this time point. | 31.6 (2.5)

4. Primary Outcome: Dosage Per Administration
Description: The median dose and range of palivizumab (milligrams) that was administered at each study visit.
Time Frame: One RSV season (5 months)
Population: as for outcome 2
Measure: Median (Full Range); unit: milligrams
Arm/Group | RSV Season 1 (S1) | RSV Season 2 (S2) | RSV Season 3 (S3) | No Matching RSV Season (NS) | Total
Number analyzed (Participants) | 39 | 45 | 32 | 4 | 120
milligrams
  V1 (S1 n=36; S2 n=44; S3 n=26; NS n=4) | 60.0 (1925.2) [40.0 to 7500.0] | 50.0 (25.8) [24.0 to 150.0] | 73.5 (26.2) [30.0 to 125.0] | 52.5 (24.2) [50.0 to 100.0] | 60.0 (1134.4) [24.0 to 7500.0]
  V2 (S1 n=32; S2 n=43; S3 n=27; NS n=0) | 77.5 (1210.7) [50.0 to 5000.0] | 70.0 (23.2) [50.0 to 150.0] | 84.0 (22.0) [43.0 to 130.0] | NA (0) [NA to NA] — No data reported for this subgroup at this time point. | 79.5 (686.0) [43.0 to 5000.0]
  V3 (S1 n=29; S2 n=42; S3 n=21; NS n=0) | 85.0 (3077.5) [60.0 to 10000.0] | 80.0 (22.7) [45.0 to 150.0] | 96.0 (21.1) [58.0 to 140.0] | NA (0) [NA to NA] — No data reported for this subgroup at this time point. | 85.5 (1795.8) [45.0 to 10000.0]
  V4 (S1 n=20; S2 n=28; S3 n=20; NS n=0) | 99.0 (1767.4) [73.0 to 8000.0] | 97.5 (285.3) [54.0 to 1600.0] | 100.0 (24.1) [65.0 to 150.0] | NA (0) [NA to NA] — No data reported for this subgroup at this time point. | 100.0 (973.1) [54.0 to 8000.0]
  V5 (S1 n=15; S2 n=13; S3 n=13; NS n=0) | 100.0 (7.8) [80.0 to 111.0] | 100.0 (18.2) [80.0 to 150.0] | 100.0 (20.1) [78.0 to 150.0] | NA (0) [NA to NA] — No data reported for this subgroup at this time point. | 100.0 [78.0 to 150.0]
  V6 (S1 n=5; S2 n=3; S3 n=2; NS n=0) | 100.0 (122) [90.0 to 123.0] | 100.0 (17.3) [100.0 to 130.0] | 101.0 (8.5) [95.0 to 107.0] | NA (0) [NA to NA] — No data reported for this subgroup at this time point. | 100.0 (12.5) [90.0 to 130.0]
  V7 (S1 n=2; S2 n=3; S3 n=0; NS n=0) | 100.0 (0) [100.0 to 100.0] | 100.0 (0) [100.0 to 100.0] | NA (0) [NA to NA] — No data reported for this subgroup at this time point. | NA (0) [NA to NA] — No data reported for this subgroup at this time point. | 100.0 (0) [100.0 to 100.0]

5. Secondary Outcome: Assessment of Pain During Injection According to Pain Scores (VAS and Modified Behavioral Pain Scale)
Description: The clinician who administered the palivizumab injection was asked to rate pain during injection using a visual analog scale (VAS) and the Modified Behavior Pain Scale (MBPS) as published by Carbajal et al., 2008. The VAS ranged from 0 (no pain) to 100 (maximum pain). The Modified Behavioral Pain Scale ranged from 0 (no pain) to 10 (maximum pain) through the evaluation of 3 items: Facial expressions, cry, and movements. If more than one injection was given at a visit, then the first injection was rated.
Time Frame: One RSV season (5 months)
Population: The analysis included participants who were administered palivizumab and had data available for the study visits listed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RSV Season 1 (S1) | RSV Season 2 (S2) | RSV Season 3 (S3) | No Matching RSV Season (NS) | Total
Number analyzed (Participants) | 39 | 45 | 32 | 4 | 120
units on a scale
  V1 VAS (S1 n=37; S2 n=43; S3 n=22; NS n=4) | 50.2 (22.3) | 64.1 (19.5) | 53.5 (25.7) | 62.5 (9.6) | 57.0 (22.3)
  V1 MBPS (S1 n=37; S2 n=43; S3 n=29; NS n=4) | 7.2 (1.7) | 7.5 (1.5) | 6.9 (1.8) | 7.8 (1.5) | 7.2 (1.7)
  V2 VAS (S1 n=33; S2 n=42; S3 n=25; NS n=0) | 55.3 (23.4) | 65.6 (18.2) | 57.2 (27.3) | NA (NA) — No data reported for this subgroup at this time point. | 60.1 (22.7)
  V2 MBPS (S1 n=34; S2 n=42; S3 n=31; NS n=0) | 7.2 (1.6) | 7.9 (1.5) | 7.3 (1.9) | NA (NA) — No data reported for this subgroup at this time point. | 7.5 (1.6)
  V3 VAS (S1 n=31; S2 n=41; S3 n=20; NS n=0) | 55.9 (23.6) | 67.8 (16.4) | 60.0 (26.6) | NA (NA) — No data reported for this subgroup at this time point. | 62.1 (21.9)
  V3 MBPS (S1 n=31; S2 n=41; S3 n=24; NS n=0) | 7.3 (1.5) | 7.9 (1.3) | 7.6 (1.8) | NA (NA) — No data reported for this subgroup at this time point. | 7.7 (1.5)
  V4 VAS (S1 n=20; S2 n=28; S3 n=19; NS n=0) | 60.3 (24.5) | 66.3 (17.1) | 62.7 (23.5) | NA (NA) — No data reported for this subgroup at this time point. | 63.5 (21.2)
  V4 MBPS (S1 n=20; S2 n=28; S3 n=22; NS n=0) | 8.2 (1.2) | 7.7 (1.4) | 7.4 (1.3) | NA (NA) — No data reported for this subgroup at this time point. | 7.7 (1.3)
  V5 VAS (S1 n=15; S2 n=13; S3 n=14; NS n=0) | 55.1 (28.1) | 65.8 (13.2) | 64.4 (27.4) | NA (NA) — No data reported for this subgroup at this time point. | 61.5 (24.1)
  V5 MBPS (S1 n=15; S2 n=13; S3 n=16; NS n=0) | 6.9 (2.1) | 7.2 (1.4) | 8.2 (1.5) | NA (NA) — No data reported for this subgroup at this time point. | 7.5 (1.8)
  V6 VAS (S1 n=5; S2 n=3; S3 n=4; NS n=0) | 51.2 (31.2) | 78.3 (2.9) | 72.0 (34.3) | NA (NA) — No data reported for this subgroup at this time point. | 64.9 (28.8)
  V6 MBPS (S1 n=5; S2 n=3; S3 n=4; NS n=0) | 7.4 (2.2) | 7.3 (0.6) | 8.8 (1.9) | NA (NA) — No data reported for this subgroup at this time point. | 7.8 (1.8)
  V7 VAS (S1 n=2; S2 n=3; S3 n=0; NS n=0) | 30.0 (0.0) | 73.3 (11.5) | NA (NA) — No data reported for this subgroup at this time point. | NA (NA) — No data reported for this subgroup at this time point. | 56.0 (25.1)
  V7 MBPS (S1 n=2; S2 n=3; S3 n=0; NS n=0) | 4.0 (1.4) | 6.7 (1.2) | NA (NA) — No data reported for this subgroup at this time point. | NA (NA) — No data reported for this subgroup at this time point. | 5.6 (1.8)

6. Secondary Outcome: Parents Knowledge of Burden of RSV Disease Via Interview by Physician
Description: An informational brochure was given to parents of participants. Parents were interviewed by the treating physician at the first study visit (V1) and last study visit (LSV) (or early termination visit [ET]) for those participants discontinuing from the study). Parental knowledge of the burden of respiratory syncytial virus (RSV) disease was assessed using a questionnaire. Parents were considered to have "good RSV awareness" if all questions were answered and at least 3 of the 4 questions regarding the burden of RSV disease were answered correctly.
Time Frame: One RSV season (5 months)
Population: The analysis included parents of participants who were administered and had data available for the study visits listed.
Measure: Number; unit: Parents of participants
Arm/Group | RSV Season 1 (S1) | RSV Season 2 (S2) | RSV Season 3 (S3) | No Matching RSV Season (NS) | Total
Number analyzed (Participants) | 39 | 45 | 32 | 4 | 120
Parents of participants
  Good RSV Awareness V1 (S1=39;S2=42;S3=32;NS=4) | 39 | 36 | 31 | 4 | 110
  Good RSV Awareness LSV (S1=28;S2=32;S3=29;NS=4) | 28 | 32 | 29 | 4 | 93
  Good RSV Awareness ET (S1=7;S2=8;S3=3;NS=0) | 7 | 7 | 3 | 0 | 17

7. Secondary Outcome: Effectiveness of Palivizumab at the End of the Observation Period is Checked by the Physician by Ranking in a Visible Analog Scale
Description: The therapeutic effect of palivizumab was assessed by the treating physician using a visual analog scale from 0 to 10, where 0 indicated that palivizumab did not match expectations at all and 10 indicated that palivizumab met all expectations. The physician rated palivizumab treatment for each participant at the last study visit (LSV) or, in the case of participants withdrawing from the study, at the early termination (ET) visit.
Time Frame: One RSV season (5 months), end of study
Population: The analysis included participants who were administered palivizumab and had data available for the study visits listed. A total of 100 participants were rated at the last study visit; 2 did not have ratings. A total of 18 participants who discontinued from the study were rated at the early termination visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RSV Season 1 (S1) | RSV Season 2 (S2) | RSV Season 3 (S3) | No Matching RSV Season (NS) | Total
Number analyzed (Participants) | 39 | 45 | 32 | 4 | 120
units on a scale
  Rating at LSV (S1 n=30;S2 n=36;S3 n=27;NS n=4) | 9.9 (0.4) | 9.8 (0.6) | 9.9 (0.5) | 10.0 (0.0) | 9.9 (0.5)
  Rating at ET visit (S1 n=7;S2 n=8;S3 n=3;NS n=0) | 10.0 (0.0) | 9.5 (0.9) | 10.0 (0.0) | NA (NA) — No participants in this subgroup were rated at an early termination visit. | 9.8 (0.6)

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the time informed consent was given until 90 days after the last dose of palivizumab. The average time from first to last study visit was approximately 125 days, with an average therapy duration of approximately 93 days.
Arm/Group | Premature Infants 33 - 35 wGA Prophylaxed With Palivizumab
Serious Adverse Events (participants affected / at risk) | 5/120
Other Adverse Events (participants affected / at risk) | 22/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Premature Infants 33 - 35 wGA Prophylaxed With Palivizumab (N=120)
Pneumonia (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Hospitalisation (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Premature Infants 33 - 35 wGA Prophylaxed With Palivizumab (N=120)
Bronchitis (Infections and infestations) | 4
Rhinitis (Infections and infestations) | 3
Varicella (Infections and infestations) | 3
Bronchitis viral (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 2
Respiratory tract infection (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.